CLINICAL TRIAL: NCT01543269
Title: A Randomized, Double Blind, Placebo Controlled Phase I Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZYT1, a Selective Thyroid Receptor (TR) ß Agonist, Following the Oral Administrations in Healthy Volunteers.
Brief Title: A Clinical Study to Evaluate the Safety,Tolerability and PK of ZYT1, Following Oral Administration in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety concerns
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYT1/1001; CTRI/2008/091/000256 (Registry Identifier: Clinical Trial Registration India)
Record Dates: First submitted 2012-02-21; First posted 2012-03-02 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Obesity; Lipid Disorders
Keywords: Obesity; Lipid disorders
MeSH Terms: conditions — Obesity; Lipid Metabolism Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ZYT1 tablets (Active Comparator): ZYT1 tablets: Route of administration: Oral Dosage: 0.5mg, 1mg, 2 mg, 4mg, 8 mg, 16mg, 32mg and 64mg
  Interventions: Drug: ZYT1
- Placebo (Placebo Comparator): Placebo tablets: Route of administration: Oral Dosage: 0.5mg, 1mg, 2 mg, 4mg, 8 mg, 16mg, 32mg and 64mg
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: ZYT1 — Oral dose of ZYT1 in fasting condition with 240±10 ml of water at sitting position in ambient temperature.
  Other Names: ZYT1 is expected to demonstrate antidyslipidemic effect and possible wt. reduction through its selective TR β agonistic activity.
  Arms: ZYT1 tablets
Drug: Placebo tablets — Oral dose of Placebo in fasting condition with 240±10 ml of water at sitting position in ambient temperature.
  Arms: Placebo

SUMMARY:
This is a clinical study to evaluate the safety, tolerability and pharmacokinetics of ZYT1, following oral administrations in healthy volunteers.

The study shall be divided into four plans as given below:

1. Plan I: Single dose escalation trial
2. Plan II: Multiple dose escalation trial
3. Plan III: Food effect trial.
4. Plan IV: Gender Effect trial.

The safety and tolerability shall be evaluated using physical examinations, Standard laboratory tests (hematology, biochemistry and urine examination), electrocardiogram (ECG) and thyroid scanning. Spontaneously reported and solicited adverse events will also be used for safety parameters.

DETAILED DESCRIPTION:
This is a clinical study to evaluate the safety, tolerability and pharmacokinetics of ZYT1, following oral administrations in healthy volunteers.

The study is divided into four plans as given below:

1. Plan I: Single dose escalation trial: A study is to evaluate safety, tolerability and PK of ZYT1 in healthy volunteers.
2. Plan II: Multiple dose escalation trial: A study is to evaluate safety, tolerability, PK and, if demonstrated, capture the Pharmacodynamics of ZYT1 in healthy volunteers.
3. Plan III: Food effect trial Effect of food on pharmacokinetics will be studied in a cross over study, with selected dose and based on limit of detection of the investigational medicinal product (IMP) in analytical methods.
4. Plan IV: Gender Effect trial . The gender effect study will be conducted after the completion of Panel S5 of single dose safety and tolerability study

The safety and tolerability shall be evaluated using physical examinations, Standard laboratory tests (hematology, biochemistry and urine examination), electrocardiogram (ECG) and thyroid scanning. Spontaneously reported and solicited adverse events will also be used for safety parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years
2. Mentally, physically and legally eligible to give informed consent.
3. Male and female volunteers weighing between 50-75kg and 45-75kg respectively.
4. Ability to communicate effectively with the study personnel.
5. Willingness to adhere to the protocol requirements.
6. Normal Thyroid Function Tests (free and total T3, free and total T4 and TSH)
7. Lipid criteria: Low density lipoprotein (LDL) cholesterol up to 160mg/dL and triglyceride (TG) level up to 500mg/dL
8. For gender effect study, only females with history of sterility or one year menopause or use of long acting nonhormonal contraceptive measures (e.g., Intra uterine device) will be recruited.

Exclusion Criteria:

1. Presence or history of hypersensitivity to any of the active or inactive ingredients of ZYT1 formulation.
2. History of thyroid disorders (any form) within 24 weeks prior to the recruitment in the study.
3. Active liver disease and/or liver transaminases greater than 1.5 X upper limit of normal (ULN).
4. Renal insufficiency (serum creatinine > 1.5mg/dL).
5. History of myocarditis, hypertrophic cardiomyopathy, valvular heart disease, restrictive cardiomyopathy, constrictive pericarditis, myocardial infarction, ischemic heart disease, stroke, congestive heart failure, cardiac arrhythmia or coronary revascularization procedure at any time.
6. Subject who has corrected QT interval (QTc)³ 450 (male) or 470 (female).
7. History or presence of musculoskeletal disorders (e.g., myopathies, myolysis, fractures due to osteoporosis, etc.)
8. History or presence of other systemic disorders or diseases (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement).
9. Subjects taking other hormonal therapies e.g., glucocorticoids, androgens or growth hormones.
10. Use of thyroid supplements (levothyroxine, liothyronine, etc.) or any preparation containing thyromimetic agents within 24 weeks prior to study entry.
11. History of coagulopathy or use of anticoagulants such as warfarin.
12. History or presence of chronic medications or any medications in the last 14 days.
13. History or presence of significant alcoholism or drug abuse within the past one-year.
14. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco products (more than 10 times per day).
15. Difficulty with donating blood.
16. Systolic blood pressure more than 140 mmHg and less than 100 mmHg and diastolic blood pressure more than 90 mmHg and less than 60 mmHg.
17. Pulse rate less than 60/minute and more than 100/minute.
18. Any clinically significant abnormal X-ray or laboratory findings during screening.
19. History or presence of any clinically significant ECG abnormalities during screening.
20. Major illness and/or Major surgery in last 3 months.
21. Volunteers who have participated in any drug research study other than the present trial within past 3 months.
22. Volunteers who have donated one unit (350ml) of blood in the past 3 months.
23. For gender effect study, female volunteers with following criteria will not be recruited:

    * History of pregnancy or lactation in the past 3 months b- Fertile female volunteers not protected against pregnancy by adequate long-term anti- fertility device or history of less than one year of menopause
    * Using hormonal contraceptives
    * Using hormone replacement therapy
    * Unable to give assurance for protection against pregnancy for 3 months after the participation in this trial
    * History of osteoporosis or history of fracture in the past 6 months
    * Positive urine pregnancy test on the day of check-in.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ZYT1 (Plan I-IV) | 14 Days
  Safety and tolerability for Plan I, II,III and IV (Time Frame upto 14 days) The safety and tolerability shall be evaluated using physical examinations, Standard laboratory tests (hematology, biochemistry and urine examination), electrocardiogram (ECG) and thyroid scanning. Spontaneously reported and solicited adverse events will also be used for safety parameters.
  Safety will be assessed by noting the number of subjects who will develop Adverse Event (AE) along with severity and causality assessment.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) (Plan I, II, III, IV) and pharmacodynamics (PD)(Plan II) | 14 days
  PK parameters:
  Plan I, III, IV:Cmax, Tmax, Area Under the Curve (AUC)0-t, AUC 0-inf, T1/2, λz, Clearance (CL), Vd Plan II:Cmin, Tmin, Cavg, % Fluctuation, Accumulation Index, Clss, Cmax, volume of distribution (VZ) or Vss For urine data (Plan I, II, III, IV):Amount recovered, recovered
  PD Parameters assessed include Bld glucose, TG, Total Chol., HDL, LDL, very low-density lipoprotein (VLDL), free fatty acid (FFA), Lipoprotein (a), Wt reduction, if any, after Plan II.
  Values compared for pre Rx and post Rx levels. PD Analysis made for differences among Rx groups as well as comparing Rx group with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Rajendrakumar H Jani, PhD(Medical), Study Director — Zydus Research Centre, Cadila Healthcare Limited,Moriya, Ahmedabad-382213, Gujrat, India
Locations (1):
- Zydus Research Centre, Cadila Healthcare Limited, Ahmedabad, Gujarat, India